CLINICAL TRIAL: NCT00505804
Title: A Randomised Open Label Pilot Study of the Efficacy of Dexmedetomidine and Haloperidol in Ventilated Patients With ICU-associated Agitation and Delirium
Brief Title: A Comparison of Dexmedetomidine and Haloperidol in Patients With Intensive Care Unit (ICU)-Associated Agitation and Delirium
Acronym: Dex
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Austin Health (Other Government)
Collaborators: The Alfred (Other)
Responsible Party: Principal Investigator, Rinaldo Bellomo, Prof, Austin Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H2004/02026
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Delirium; Agitation; Ventilator Weaning; Respiration, Artificial; Intensive Care
Keywords: dexmedetomidine; haloperidol
MeSH Terms: conditions — Delirium; Psychomotor Agitation; Respiratory Aspiration | interventions — Dexmedetomidine; Haloperidol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: dexmedetomidine
- 2 (Active Comparator)
  Interventions: Drug: haloperidol

INTERVENTIONS:
Drug: dexmedetomidine — Dexmedetomidine IV infusion of 0.0 to 0.7 mg/kg/min for as long a deemed necessary by the treating clinician.
  Arms: 1
Drug: haloperidol — Haloperidol IV loading dose of 2.5mg, followed by a continuous infusion of 0.0 to 2mg/hr for as long as deemed necessary by the treating clinician
  Arms: 2

SUMMARY:
The purpose of the study is to determine whether dexmedetomidine is a more effective medication than haloperidol in the treatment of agitation and delirium in patients receiving mechanical ventilation in an intensive care unit. Haloperidol is a medication conventionally used for this purpose.

The investigators will study only patients who have recovered from their illness to the point that, were it not for agitation and delirium, they would no longer require mechanical ventilation.

The investigators hypothesize that patients receiving dexmedetomidine will be able to discontinue mechanical ventilation earlier than those receiving haloperidol.

DETAILED DESCRIPTION:
Up to 80% of patients undergoing intensive care have delirium. Early in the ICU stay, delirium and agitation are usually prevented using analgesic and sedative drugs which essentially render the patient unconscious. This is appropriate in the context of aggressive treatment of pathophysiological instability, which often requires multiple painful procedures. However, after the underlying pathophysiological problem has resolved, patients sometimes remain delirious and agitated. This often requires ongoing heavy sedation, which in turn necessitates continued mechanical ventilation, and can worsen the (temporarily masked) delirium. Prolonged mechanical ventilation increases the risk of ventilator associated pneumonia and other life threatening complications.

The drug most commonly used to treat delirium is haloperidol, which reduces hallucinations and unstructured thought patterns, but also reduces the interaction with the environment. Haloperidol has significant side effects, including extrapyramidal reactions (in 1-10% of patients), neuroleptic malignant syndrome (in which it is the cause in 50% of cases), and prolonged QT syndrome (which can precipitate fatal arrhythmias).

An ideal sedative agent in this context would have fewer side effects, relieve agitation without causing excessive sedation, and be easily titrated. An analgesic action might allow less opioid use, also lessening delirium. Early studies in other contexts suggest dexmedetomidine has all these properties.

The investigators hypothesise that patients with ICU-associated delirium after the resolution of their underlying pathological process who receive dexmedetomidine will be able to be extubated earlier than those who receive haloperidol.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible for the study if, in the opinion of the treating clinician, they continue to require mechanical ventilation only because their degree of agitation requires such a high dose of sedative medication (midazolam or propofol, the only commonly used specific sedatives in our unit) that extubation is not possible.

Exclusion Criteria:

* Patients who could not be extubated even if delirium or agitation were corrected. This will include:

  * Patients receiving high dose opioid analgesia (>20 m/morphine/day)
  * Patients shortly to return to the operating theatre
  * Patients undergoing repeated invasive procedures, in whom it is desirable to maintain deep sedation.
  * Patients likely to require ongoing airway protection or control, or ventilatory support (for example, spinal patients with an inadequate vital capacity)
* Known allergy to haloperidol or alpha2 agonists

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-01; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Time from the commencement of treatment to extubation | days
  the tiem taken to extubate the patient

SECONDARY OUTCOMES:
Time taken to achieve a satisfactory sedation score (score 3 or 4 on the Riker scale) | hours
  time to sedation score
The need for supplemental sedative and analgesic medication (morphine, midazolam or propofol, as clinically indicated) | During delivery of trial medication
Average Riker score for agitation | During delivery of trial medication
Average RASS score for agitation | During delivery of trial medication
Need for re-intubation | During the same ICU admission
Average Bergeron ICDSC score for delirium | During delivery of trial medication
Duration of ICU stay | days

CONTACTS AND LOCATIONS:
Overall Officials: Rinaldo Bellomo, MD FJFICM, Principal Investigator — Austin Health, University of Melbourne; Michael C Reade, MBBS FJFICM, Study Director — Austin Health, University of Melbourne

REFERENCES:
- [Derived] Reade MC, O'Sullivan K, Bates S, Goldsmith D, Ainslie WR, Bellomo R. Dexmedetomidine vs. haloperidol in delirious, agitated, intubated patients: a randomised open-label trial. Crit Care. 2009;13(3):R75. doi: 10.1186/cc7890. Epub 2009 May 19. PMID 19454032